CLINICAL TRIAL: NCT00478660
Title: Review of Safety and Efficacy With Adalimumab in Patients With Active Ankylosing Spondylitis - An Open-Label Study to Evaluate the Response to Adalimumab in Patients Who Have Failed Standard Therapy or TNF-Alpha Inhibitors (RHAPSODY)
Brief Title: An Open-Label Study to Evaluate the Response to Adalimumab in Patients With Active Ankylosing Spondylitis Who Have Failed Standard Therapy or TNF-Alpha Inhibitors (RHAPSODY)
Acronym: RHAPSODY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: M05-760
Record Dates: First submitted 2007-05-23; First posted 2007-05-25 (Estimated); Last update posted 2007-10-10 (Estimated); Status verified 2007-10

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Adalimumab

INTERVENTIONS:
Drug: adalimumab (Humira)

SUMMARY:
Due to the rigor of the clinical development program of adalimumab for the indication of AS, the population of subjects with active AS that could enroll in previous phase 3 studies was limited. Therefore, it is necessary to further evaluate the use of adalimumab in a setting that mimics day-to-day clinical practice to obtain further safety and efficacy data by allowing subjects meeting the characteristics noted below to enter this study:

* Subjects who failed another TNF inhibitor (etanercept, infliximab)
* Subjects with advanced spinal ankylosis
* Subjects with AS associated disorders (i.e., uveitis, IBD, and psoriasis)

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent and to comply with the requirements of the study protocol
* Males and females 18 years of age or older
* Diagnosis of AS according to the modified New York Criteria for Ankylosing Spondylitis 1984.24
* Documented active AS based on the opinion of a physician for at least 3 months
* Active AS with BASDAI >= 4 at the Screening Visit
* Unsatisfactory response to standard AS therapies in accordance with the current national guidelines for treatment of AS with TNF inhibitors (if applicable) including a minimum of failing at least one NSAID. National guidelines (if applicable) must be followed if the guidelines are more strict regarding the use of TNF inhibitors for the treatment of AS
* Use of reliable method of contraception, e.g., IUDs, condoms, or hormone (oral, implantable, or injectable) contraceptives by all female subjects of childbearing potential. Subject must follow the manufacture's recommendations of contraception prior to the administration of study drug and through 150 days following the last administration of adalimumab
* Able and willing to self-administer sc injections or have available a suitable person to administer sc injections
* A negative pregnancy test (serum HCG) for women of childbearing potential prior to start of study treatment
* Subject must be evaluated for active and latent TB infection by using a PPD skin test, T SPOT-TB test, chest x-ray and a detailed review of the subject's medical history. Guidelines regarding the treatment of latent TB must be followed prior to the administration of adalimumab

Exclusion Criteria:

* Prior treatment with any investigational agent within 30 days, or five half-lives of the product, which ever is longer
* Treatment within the last six weeks with infliximab or within the last three weeks with etanercept or previous treatment at any time with adalimumab
* Known allergy to excipients of adalimumab formulation
* History of or current acute inflammatory joint disease of origin other than AS, e.g., rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus etc
* Treatment with corticosteroids (prednisolone equivalents) under the following conditions:

  * Dose is >10 mg/d systemically within the 28 days before screening
  * Intraarticular injections or infiltrations of peripheral joints and tendons within 28 days before or at screening
  * Intraarticular injections of sacroiliac joints without therapeutic response <=14 days before screening
* Other medical conditions: uncontrolled diabetes, unstable ischemic heart disease, congestive heart failure (NYHA III-IV), recent stroke (within three months), chronic leg ulcer and any other condition (e.g., indwelling urinary catheter) which, in the opinion of the investigator, would put the subject at risk by participation in the study
* History of cancer or malignant lymphoproliferative disease other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix
* History of positive serology for hepatitis B indicating active infection or history of positive serology for hepatitis C
* History of positive HIV status
* Persistent or recurrent infections or severe infections requiring hospitalization or treatment with iv antibiotics within 30 days, or oral antibiotics within 14 days prior to enrollment
* Previous diagnosis or signs highly indicative of central nervous system demyelinating diseases (e.g., optic neuritis, ataxia, apraxia)
* History of active tuberculosis, histoplasmosis or listeriosis
* Female subjects who are pregnant or breast-feeding
* History of clinically significant drug or alcohol abuse in the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1250 (Actual)
Dates: Start 2006-02

PRIMARY OUTCOMES:
ASAS 20/40/50/70
ASAS 5/6
BASDAI score

SECONDARY OUTCOMES:
Adverse events
Laboratory data
Vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Paperiello, Study Director — Abbott
Locations (171):
- Austria (3):
  - Graz
  - Innsbruck
  - Vienna
- Belgium (9):
  - Aalst
  - Belsele
  - Bruges
  - Charleroi
  - Erembodegem
  - Genk
  - Ghent
  - Hasselt
  - Ostend
- Denmark (5):
  - Frederiksberg
  - Holstebro
  - Kolding
  - Randers
  - Silkeborg
- Finland (4):
  - Helsinki
  - Hyvinkää
  - Kouvola
  - Turku
- France (44):
  - Aix-en-Provence
  - Aix-les-Bains
  - Amiens
  - Angers
  - Belfort
  - Berck
  - Besançon
  - Bordeaux
  - Boulogne-Billancourt
  - Brest
  - Caen
  - Cahors
  - Clermont-Ferrand
  - Corbeil-Essonnes
  - Créteil
  - Dijon
  - Grenoble
  - Le Kremlin-Bicêtre
  - Le Mans
  - Libourne
  - Liévin
  - Lille
  - Limoges
  - Lomme
  - Lyon
  - Marseille
  - Montivilliers
  - Montpellier
  - Mulhouse
  - Nantes
  - Nice
  - Orléans
  - Paris
  - Pau
  - Poitiers
  - Reims
  - Rennes
  - Saint-Brieuc
  - Saint-Etienne
  - Strasbourg
  - Toulouse
  - Tours
  - Valenciennes
  - Vandœuvre-lès-Nancy
- Germany (43):
  - Bad
  - Bad Bentheim
  - Bad Bramstedt
  - Bad Nauheim
  - Berlin
  - Chemnitz
  - Cologne
  - Cottbus
  - Damp
  - Dresden
  - Duisburg
  - Düsseldorf
  - Erfurt
  - Erlangen
  - Frankfurt
  - Freiburg im Breisgau
  - Goslar
  - Göttingen
  - Hamburg
  - Hanover
  - Heidelberg
  - Herne
  - Hildesheim
  - Hofheim
  - Hoyerswerda
  - Jena
  - Kiel
  - Leipzig
  - München
  - Neubrandenburg
  - Osnabrück
  - Planegg
  - Ratingen
  - Regensburg
  - Rostock
  - Sendenhorst
  - Stuttgart
  - Tübingen
  - Villingen
  - Vogelsang/Gommern
  - Würzburg
  - Zerbst
  - Zeven
- Greece (6):
  - Athens
  - Heraklion
  - Ioannina
  - Larissa
  - Pátrai
  - Thessaloniki
- Ireland (2):
  - Cork
  - Dublin
- Italy (7):
  - Florence
  - Monserrato
  - Napoli
  - Palermo
  - Potenza
  - Reggio Emilia
  - Roma
- Netherlands (5):
  - Den Helder
  - Enschede
  - Flushing
  - Leeuwarden
  - Zwolle
- Norway (5):
  - Haugesund
  - Levanger
  - Lillehammer
  - Tromsø
  - Trondheim
- Spain (14):
  - A Coruña
  - Alicante
  - Asturias
  - Barakaldo
  - Barcelona
  - Burgos
  - Las Palmas de Gran Canaria
  - Madrid
  - Pamplona
  - Valencia
  - Valladolid
  - Vitoria-Gasteiz
  - Vizcaya
  - Zaragoza
- Sweden (4):
  - Eskilstuna
  - Örebro
  - Östersund
  - Vaxjo
- Switzerland (2):
  - Bern
  - Zurich
- United Kingdom (18):
  - Aberdeen
  - Avon
  - Birmingham
  - Cambridge
  - Greater Manchester
  - Harrow
  - Huddersfield
  - Leeds
  - Liverpool
  - London
  - Merseyside
  - Newcastle upon Tyne
  - Oxford
  - Portsmouth
  - Sheffield
  - Southampton
  - Truro
  - Wigan

REFERENCES:
- [Derived] Rudwaleit M, Van den Bosch F, Kron M, Kary S, Kupper H. Effectiveness and safety of adalimumab in patients with ankylosing spondylitis or psoriatic arthritis and history of anti-tumor necrosis factor therapy. Arthritis Res Ther. 2010;12(3):R117. doi: 10.1186/ar3054. Epub 2010 Jun 16. PMID 20553600
- [Derived] Rudwaleit M, Claudepierre P, Kron M, Kary S, Wong R, Kupper H. Effectiveness of adalimumab in treating patients with ankylosing spondylitis associated with enthesitis and peripheral arthritis. Arthritis Res Ther. 2010;12(2):R43. doi: 10.1186/ar2953. Epub 2010 Mar 15. PMID 20230622
- [Derived] Rudwaleit M, Claudepierre P, Wordsworth P, Cortina EL, Sieper J, Kron M, Carcereri-De-Prati R, Kupper H, Kary S. Effectiveness, safety, and predictors of good clinical response in 1250 patients treated with adalimumab for active ankylosing spondylitis. J Rheumatol. 2009 Apr;36(4):801-8. doi: 10.3899/jrheum.081048. Epub 2009 Feb 27. PMID 19273449
- [Derived] Rudwaleit M, Rodevand E, Holck P, Vanhoof J, Kron M, Kary S, Kupper H. Adalimumab effectively reduces the rate of anterior uveitis flares in patients with active ankylosing spondylitis: results of a prospective open-label study. Ann Rheum Dis. 2009 May;68(5):696-701. doi: 10.1136/ard.2008.092585. Epub 2008 Jul 28. PMID 18662932